CLINICAL TRIAL: NCT01614717
Title: Triple Chamber Pacing in HOCM Patients - TRICHAMPION STUDY
Brief Title: Triple Chamber Pacing in Hypertrophic Obstructive Cardiomyopathy (HOCM) Patients - TRICHAMPION STUDY
Acronym: TRICHAMPION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-11-030-EU-HF
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Hypertrophic Cardiomyopathy With Obstruction
Keywords: Hypertrophic Obstructive Cardiomyopathy; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): CRT-P Implant. Patients randomized in Treatment Group will have the device programmed to optimized DDD pacing
  Interventions: Device: CRT-P Implant
- Control Group (Placebo Comparator): CRT-P Implant. Patients randomized in the control Group will have the device programmed to back-up pacing AAI
  Interventions: Device: CRT-P Implant

INTERVENTIONS:
Device: CRT-P Implant — All patients will be implanted with a CRT-P device, then randomized to Treatment or Control Group

SUMMARY:
This investigation is a prospective, randomized, single-blinded and multicenter design.

The purpose of this study is to evaluate the benefit of atrial-synchronous biventricular (BiV) pacing in severely symptomatic hypertrophic obstructive cardiomyopathy (HOCM) patients with severe Left Ventricular Outflow Tract (LVOT) obstruction implanted with a Cardiac Resynchronization Therapy - Pacing (CRT-P) device.

Randomization

* Implant will be performed (CRT-P).
* Patients will be randomized 1:1 to either Treatment Group (Optimized Biventricular (DDD) pacing) or Control Group (Back-up Atrial (AAI) pacing) during the first 12 months:
* Treatment Group. The patient´s device is programmed to optimized DDD BiV pacing
* Control Group. The patient´s device is programmed to back-up pacing AAI.
* After 12 months, the patients initially randomized to the Treatment Group (Optimized DDD Pacing) will continue in the same group. The patients initially randomized to Control Group (AAI Back-up Pacing) will be changed to the Treatment Group (Optimized DDD Pacing). And all the patients will be followed 12 months more.

DETAILED DESCRIPTION:
Data collection

* In clinic Follow ups (FU): Enrollment, Baseline, Implant, Pre-discharge, 3 months (M), 12 M, 15 M and 24 M.
* Phone call FU: 6 M, 9 M, 18 M and 21 M.

ELIGIBILITY:
Inclusion Criteria:

1. Unequivocal diagnosis of hypertrophic cardiomyopathy (HCM), on the basis of 2-dimensional echocardiographic demonstration of a hypertrophied (wall thickness ≥15 mm) and nondilated Left Ventricle (Left Ventricle End Diastolic Diameter (LVEDD) < 55mm) confirmed by a Core Lab Echo (Appendix I).
2. Significant resting (not provoked) LV outflow tract obstruction, on the basis of peak LVOT gradient ≥50 mmHg, estimated by continuous wave Doppler and confirmed by a Core Lab Echo (Appendix I).
3. Presence of refractory symptoms (exertional dyspnea or chest pain) despite of optimal treatment with betablockers and/or verapamil for at least 3 months (NYHA class >II).
4. Patients that refuse or have contraindication for septal myectomy or septal ablation (i.e., comorbidity, inappropriate coronary anatomy for septal ablation), that prefer cardiac pacing, or that are at high risk for developing heart block following septal myectomy or septal ablation.

6. Patient's age is 18 years or greater. 7. Patients must indicate their understanding of the study and willingness to participate by signing the appropriate informed consent form.

8. Patients must be willing and able to comply with all study requirements.

Exclusion Criteria:

1. Known causes of cardiac hypertrophy as infiltrative cardiomyopathy, aortic stenosis and severe uncontrolled hypertension.
2. Permanent or persistent atrial fibrillation.
3. Previous septal myectomy or septal ablation.
4. Any indication for permanent pacing, except for HOCM.
5. Any indication for an Implantable Cardioverter Defibrillator (ICD).
6. Systemic disease that would preclude completion of the protocol.
7. Any disability or limitations to correctly understand or complete the study (physical, intellectual, logistical).
8. Patients with a life expectancy <24 months (based on investigator assessment).
9. Patients who are or may potentially be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the percentage of HOCM patients with severe LVOT obstruction implanted with a CRT-P device that have symptomatic improvement at 12 months. | 12 months
  The primary endpoint of the study is to evaluate the percentage of HOCM patients with severe LVOT obstruction implanted with a CRT-P device that have symptomatic improvement at 12 months post-implant.
  The symptomatic improvement is a combined endpoint defined as:
  * An improvement of at least one New Yorl Heart Association (NYHA) functional class and
  * An improvement of 10 points in the Quality of Life (QoL) Questionnaire score and
  * An increase >10% in bike exercise time in the steady state Cardiopulmonary Exercise Test (CPET).

CONTACTS AND LOCATIONS:
Overall Officials: Josep Brugada, Proffesor, Principal Investigator — Hospital Clinic I Provincial, Barcelona, Spain; Antonio Berruezo, Dr., Principal Investigator — Hospital Clinic I Provincial, Barcelona, Spain
Locations (1):
- Hospital Universitario Clinic I Provincial, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No